CLINICAL TRIAL: NCT00301587
Title: A Randomized, Double-Blind, Two-Part, Parallel-Group, Comparative Study to Evaluate Blood Folate Levels in Women Taking an Oral Contraceptive With and Without Folic Acid
Brief Title: A Study to Evaluate Folate Levels in Women Taking Oral Contraceptives
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision to not fund further development of women's health new drug development programs.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002377
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2011-07

CONDITIONS: Neural Tube Defects; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Nervous System Malformations
Keywords: spina bifida; birth defects; folic acid; nervous system diseases; folate; Vitamin B
MeSH Terms: conditions — Neural Tube Defects; Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Nervous System Malformations; Spinal Dysraphism; Congenital Abnormalities; Nervous System Diseases | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Norgestimate-ethinyl estradiol, with or without folic acid

SUMMARY:
The purpose of this study is to compare red blood cell folate levels in women who are taking oral contraceptives with or without folic acid

DETAILED DESCRIPTION:
Studies have shown an association between increased folic acid (a synthetic form of folate, a B-vitamin) intake and reduction of a birth defect referred to as neural tube defects (NTDs). If women using contraception were to receive a combination of an oral contraceptive and folic acid, they may have the benefit of increased blood folate levels, which could reduce the risk of NTDs. This is a multi-center, double-blind study designed to study red blood cell folate levels in women who are taking oral contraceptives with or without folic acid. Patients will receive oral contraceptives with or without folic acid for 8 cycles of 28 days each. The study will consist of 2 parts of 4 cycles each. All patients will receive oral contraceptives throughout both parts of the study, patients may or may not receive folic acid in combination with the oral contraceptive during 1 or both parts of the study. The concentration of red blood cell folate will be determined by laboratory tests after Cycles 1, 2, 4, 5, 6 and 8. Safety evaluations (incidence of adverse events, electrocardiograms, physical examinations, laboratory tests) will be performed throughout the study. Patients may also participate in an optional portion of the study in which their genetic material is analyzed to see if contains something that would affect the way folic acid is used by their bodies. The study hypothesis is that women taking an oral contraceptive with folic acid will have increased levels of red blood cell folate compared to women taking an oral contraceptive without folic acid. Some women who receive the oral contraceptive with folic acid during the first four cycles will be transitioned to an oral contraceptive without folic acid for Cycles 5-8. In this group of women, the rate of decrease in red blood cell folate levels will be measured. Norgestimate 250 micrograms (mcg)-ethinyl estradiol 35 mcg tablets, with or without folic acid 400 mcg, 2 tablets taken by mouth daily between 6:00 a.m. and 10:00 a.m. for 8 cycles of 28 days duration each for a total of 224 days

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant post menarcheal, premenopausal females who agree to use the assigned study medication as contraception during the study
* Non-vegan
* Non-smoker or no history of tobacco use within 6 months
* Willing to follow protocol-specific prohibitions and restrictions regarding diet, smoking and use of other medications

Exclusion Criteria:

* Have taken multivitamins, folic-acid containing supplements, or highly fortified (i.e., >200 mcg folic acid/serving) cereals within 30 days of entry in to the study
* history or presence of blood clots in the veins, strokes or other blood clotting disorder, liver tumor from pervious contraceptive or estrogen use, disease of the blood vessels of the brain or heart disease, uncontrolled high blood pressure, cancer in any part of the body, diabetes mellitus with complications in the flow of blood in the body, jaundice, visual disturbance, liver disease, undiagnosed vaginal bleeding, gastric bypass surgery, ulcerative colitis or other digestive system disorders, abnormal thyroid function, Vitamin B 12 deficiency or very high red blood cell folate levels, alcohol or substance abuse, positive for drugs of abuse
* recent use of hormonal contraceptives
* on any weight reduction diet
* blood donation within 30 days of study entry

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2004-12 (Estimated)

PRIMARY OUTCOMES:
Part 1: Change in concentration of folate in red blood cells (RBC) from the start of the study to Cycle 4 (4 cycles of 28 days of treatment)

SECONDARY OUTCOMES:
Change in plasma folate concentration from baseline to Cycle 4; Levels and change from baseline in RBC and plasma folate concentration at specified time points during the study including Cycles 1, 2, 4, 5, 6, 8

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.